CLINICAL TRIAL: NCT01192217
Title: A Prospective Randomized Study of a Modified Two-port Thoracoscopic Technique Versus Axillary Minithoracotomy for the Treatment of Recurrent Spontaneous Pneumothorax.
Brief Title: Video-assisted Thoracic Surgery (VATS) Versus Axillary Mini-thoracotomy for the Treatment of Recurrent Spontaneous Pneumothorax
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AHEPA University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AHEPACTS-01
Record Dates: First submitted 2010-08-27; First posted 2010-09-01 (Estimated); Last update posted 2010-09-01 (Estimated); Status verified 2009-01

CONDITIONS: Pneumothorax
Keywords: video-assisted thoracic surgery; axillary mini-thoracotomy; bullectomy
MeSH Terms: conditions — Pneumothorax | interventions — Thoracic Surgery, Video-Assisted; Thoracotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- VATS group (Active Comparator)
  Interventions: Procedure: Modified thoracoscopic technique
- Mini-thoracotomy group (Active Comparator)
  Interventions: Procedure: Axillary mini-thoracotomy

INTERVENTIONS:
Procedure: Modified thoracoscopic technique — Two-port thoracoscopic technique
  Other Names: VATS
  Arms: VATS group
Procedure: Axillary mini-thoracotomy — Axillary mini-thoracotomy
  Other Names: Thoracotomy
  Arms: Mini-thoracotomy group

SUMMARY:
The investigators conducted a prospective randomized study to compare axillary minithoracotomy versus a modified two-port thoracoscopic technique for surgical pleurodesis in patients with recurrent spontaneous pneumothorax operated in a single institution.

The main objective of the study was to investigate possible differences regarding short- and long-term clinical outcome between the two different techniques.

ELIGIBILITY:
Inclusion Criteria:

* ipsilateral recurrent spontaneous pneumothorax
* first episode of contralateral pneumothorax

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2006-01; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
pneumothorax recurrence rate
  Recurrence rate
Postoperative complication rate
  Postoperative complications
Patient satisfaction with treatment

SECONDARY OUTCOMES:
Duration of one-lung ventilation
Total operative time
Duration of chest tube drainage
Length of postoperative hospital stay
Incidence of chronic pain

CONTACTS AND LOCATIONS:
Overall Officials: Christos Papakonstantinou, Professor, Study Chair — AHEPA University Hospital
Locations (1):
- AHEPA University Hospital Department of Cardiothoracic Surgery, Thessaloniki, Greece